CLINICAL TRIAL: NCT05616364
Title: Comparison of the Efficacy of Intravenous Dexmedetomidine and Tramadol in Control of Post Spinal Shivering in Obstetric Patients Undergoing Lower Segment Cesarean Section
Brief Title: Compair Efficacy of iv Dexmedetomidine & Tramadol for Post Spinal Shivering in Obs Patients Undergoing Cesarean Section
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sana Bahadur (Other Government)
Responsible Party: Sponsor-Investigator, Sana Bahadur, Dr.Sana bahadur, Sheikh Zayed Medical College
Organization: Sheikh Zayed Medical College (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sheikh Zayed Medical College &
Record Dates: First submitted 2022-10-09; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Post Spinal Shivering
MeSH Terms: interventions — Dexmedetomidine; Tramadol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine is a sedative, analgesic, anxiolytic, sympatholytic, and opioid-sparing alpha 2 adrenergic agonist with good selectivity and specificity.It has been shown to lower the threshold for shivering. Dexmedetomidine does not affect the locus ceruleus of the spinal cord, and it does not cause respiratory depression. [8] In postoperative patients, dexmedetomidine lowers cortisol and norepinephrine levels, as well as blood glucose, interleukin (IL)-6, tumour necrosis factor-a, and C-reactive protein, and raises interleukin-10. Moreover, because Dexmedetomidine does not affect upper airway reflexes, it is an excellent option.It was believed that the sedative impact of intravenous injection on newborn infants was very minimal and could be disregarded due to the delayed sedative effects
  Interventions: Drug: Dexmedetomidine injection
- Tramadol (Experimental): Tramadol, a centrally acting analgesic with -opioid agonist properties and little action on kappa and delta receptors, has been proven to be beneficial in preventing post-spinal shivering. The method of action is thought to be through a modulatory influence on central monoaminergic pathways, which inhibits noradrenaline and serotonin neuronal absorption in the spinal cord while boosting hydroxyltryptamine production, resetting the body temperature regulatory center. [3] However, it has many side effects, including nausea, vomiting, and dizziness, which add to the patient's pain. [5] Hence research into novel solutions with adequate safety and effectiveness is strongly advised. In this sense, despite taking into account the gold standard for post spinal shivering control is pethidine. it is contraindicated in breastfeeding which is both legally and ethically challenging for women.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Dexmedetomidine injection — Dexmedetomidine intravenous
  Arms: Dexmedetomidine
Drug: Tramadol — Tramadol intravenous
  Arms: Tramadol

SUMMARY:
When opposed to GA,SA is recommended during c section. Shivering is more prevalent and inconvenient complication of spinal anaesthesia, with 40 to 70% incidence rate. Tramadol has been proven to be beneficial in preventing post spinal shivering. Dexmedetomidine is a sedative, analgesic, anxiolytic, sympatholytic and opioid-sparing alpha adrenergic agonist. It has been shown to lower the threshold for shivering. The study aims to search for best drug for blunting shivering response.

DETAILED DESCRIPTION:
When opposed to general anaesthesia (GA), spinal anaesthesia (SA) is recommended during caesarean section (CS) because of various advantages, including the prevention of GA-related neurotoxicity, its early onset and ease of administration, and the reduction of post-operative pain. Intraoperative shivering is the most prevalent irritating and inconvenient complication of spinal anaesthesia, and it is a very distressing experience that causes physiological stress to both patients and perioperative physicians and operating surgeons. Shivering is a skeletal muscular movement that occurs involuntarily and repeatedly. It's a common post-anesthesia adverse effect, with a 40-70% incidence rate.Shivering is not only physically unpleasant for the sufferer, but it can also have several negative consequences. It can cause pain, and discomfort for patients, obstruct monitoring techniques, raise intraocular and intracranial pressures, and double or even triple oxygen and carbon dioxide intake.Various pharmacological and non-pharmacological strategies for managing intraoperative shivering are discussed.

Tramadol, a centrally acting analgesic with -opioid agonist properties and little action on kappa and delta receptors, has been proven to be beneficial in preventing post-spinal shivering. The method of action is thought to be through a modulatory influence on central monoaminergic pathways, which inhibits noradrenaline and serotonin neuronal absorption in the spinal cord while boosting hydroxyltryptamine production, resetting the body temperature regulatory center.However, it has many side effects, including nausea, vomiting, and dizziness, which add to the patient's pain. Hence research into novel solutions with adequate safety and effectiveness is strongly advised. In this sense, despite taking into account the gold standard for post spinal shivering control is pethidine. it is contraindicated in breastfeeding which is both legally and ethically challenging for women.

Dexmedetomidine is a sedative, analgesic, anxiolytic, sympatholytic, and opioid-sparing alpha 2 adrenergic agonist with good selectivity and specificity.It has been shown to lower the threshold for shivering.Dexmedetomidine does not affect the locus ceruleus of the spinal cord, and it does not cause respiratory depression. In postoperative patients, dexmedetomidine lowers cortisol and norepinephrine levels, as well as blood glucose, interleukin (IL)-6, tumour necrosis factor-a, and C-reactive protein, and raises interleukin-10. Moreover, because Dexmedetomidine does not affect upper airway reflexes, it is an excellent option.It was believed that the sedative impact of intravenous injection on newborn infants was very minimal and could be disregarded due to the delayed sedative effects.

These drugs have well-defined roles to blunt the "shivering response" and hence have been used in different comparative studies to develop the single best drug of choice. Yet, there is no consensus over a single drug. In our research, we intend to compare IV Tramadol and IV Dexmedetomidine for controlling post spinal shivering in obstetric patients. The study aims to search for the best drug for blunting the shivering response, which may prove fatal in any patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient who will give consent
* ASA 2 patients
* Female gender of age 18 to 38

Exclusion Criteria:

* Patient allergic to any drugs
* Uncontrolled HTN
* Antepartum
* Cardiomyopathy
* Peripartum haemorrhage
* Eclampsia
* Patients refuse to give consent

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of post spinal shivering by observing grades of shivering | 10 minutes
  Control of post spinal shivering Dexmedetomidine and tramadol for post spinal shivering